CLINICAL TRIAL: NCT00471614
Title: Uridine Supplementation, Mitochondrial Function, and Glucose Metabolism in HIV
Brief Title: Effects of Uridine Supplementation on Metabolic Side Effects of Stavudine and Zidovudine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Morris Schambelan, Emeritus Professor of Medicine, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT003374-01A1 (NIH)
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections; Insulin Resistance; Hyperlactatemia
Keywords: HIV; AIDS; uridine; mitochondria; insulin resistance; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Insulin Resistance; Hyperlactatemia; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): NucleomaxX
  Interventions: Drug: NucleomaxX (contains uridine)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: NucleomaxX (contains uridine)

INTERVENTIONS:
Drug: NucleomaxX (contains uridine) — Escalated doses of NucleomaxX tid

SUMMARY:
The purpose of this study is to determine whether uridine supplementation will improve insulin sensitivity and overall carbohydrate metabolism in HIV-positive subjects who are currently undergoing treatment with antiretroviral regimens containing stavudine or zidovudine and who have evidence of impaired mitochondrial function and insulin resistance.

DETAILED DESCRIPTION:
Treatment of HIV infection with nucleoside analogue reverse transcriptase inhibitors (NRTIs) has been associated with numerous toxicities that have been attributed to impaired mitochondrial function secondary to a reduction in the levels of mitochondrial DNA (mtDNA). Abnormalities in mitochondrial function have been implicated in the development of insulin resistance in patients with HIV infection and have also been hypothesized to underlie many of the pathophysiologic features of type 2 diabetes mellitus in non-HIV infected individuals.

Uridine, a pyrimidine nucleoside that plays an essential role in the synthesis of RNA and other key physiologic processes, has been proposed as a therapy for NRTI-induced mitochondrial dysfunction. Uridine supplementation protected bone marrow cells from the toxicity of zidovudine, normalized the growth of neurons exposed to NRTIs, and abrogated mitochondrial toxicity of NRTIs in HepG2 cells in vitro. A food supplement called NucleomaxX®, extracted from the stem of sugar cane, raises plasma uridine concentrations to levels known to prevent mitochondrial toxicity in vitro. In a recent case report, oral administration of uridine, given in the form of NucleomaxX®, ameliorated the mitochondrial toxicity caused by stavudine and led to improvements in myalgias and liver and muscle enzymes, despite continuing treatment with stavudine. In a clinical study of 14 HIV-infected patients treated with stavudine or zidovudine, NucleomaxX® led to improved hepatic mitochondrial function as assessed by the 13C-methionine breath test.

We will perform a randomized double-blind placebo-controlled study in 20 HIV-positive subjects who are currently undergoing treatment with antiretroviral regimens containing stavudine or zidovudine and who have evidence of impaired mitochondrial function and insulin resistance. Subjects will be hospitalized in the SFGH CTSI Clinical Research Center (CCRC) for 6 days to undergo comprehensive metabolic studies. Subjects will then be randomized, in a 1:1 fashion, to receive either NucleomaxX® or placebo for two months, after which they will repeat the 6-day CCRC-based assessments. This study is designed to test the hypothesis that, in comparison to placebo, uridine supplementation will enhance mitochondrial function, and this will be associated with concomitant improvements in glucose and lipid metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection
* HIV-1 RNA <10,000 copies/mL within 30 days of study entry
* Treatment with stavudine or zidovudine for at least 12 months prior to entry and no plan to discontinue for the duration of the study
* Stable antiretroviral regimen for at least 3 months prior to entry and no plan to change antiretroviral therapy for the duration of the study
* Mitochondrial dysfunction as evidenced by a fasting plasma lactate level > 1.5 mmol/L
* Insulin resistance as evidenced by a HOMA-IR > 2.77 as calculated from fasting blood samples (for glucose and insulin) obtained during the screening visit
* Karnofsky performance score >= 80
* Women who are on stable regimens of hormonal contraceptives or hormone replacement therapy for at least 6 months prior to enrollment may participate
* Men who are on stable doses of testosterone replacement therapy for 6 months prior to enrollment may participate
* Subjects on a stable dose of lipid lowering agents for 6 months prior to enrollment may participate

Exclusion Criteria:

* Serum creatinine and blood urea nitrogen > 1.5 upper limit of normal (ULN)
* Direct bilirubin >2 X ULN
* AST (SGOT) or ALT (SGPT) >5 x ULN
* Hgb < 8.5 g/dL
* Abnormal hepatitis B or C serology
* A clinical diagnosis of diabetes mellitus or a fasting glucose > 126 mg/dl
* Physical or functional obstruction to food intake or impaired absorption
* A clinically suspected concomitant treatable infection that has not yet been treated
* An opportunistic infection within the preceding 30 days
* Ascites
* Pregnancy
* Treatment with growth hormone, anabolic steroids (including supraphysiologic doses of testosterone), glucocorticoids, insulin, sulfonylureas, metformin, thiazolidinediones, or appetite stimulants within preceding 6 months
* Dementia, active drug or alcohol abuse or dependence, or other conditions that would preclude adherence to the protocol or the ability to provide informed consent.
* Any other condition that, in the opinion of the investigators, would put the subject at risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity as measured by euglycemic hyperinsulinemic clamp (with simultaneous stable isotope tracer studies) | 2 months

SECONDARY OUTCOMES:
Change in body composition (DEXA and CT imaging) | 2 months
Change in insulin secretion (frequently sampled intravenous glucose tolerance test) | 2 months
Change in resting energy expenditure (indirect calorimetry) | 2 months
Change in markers of oxidative stress | 2 months
Change in mtDNA levels (measured in muscle biopsy) | 2 months
Change in HIV disease markers | 2 months
Adverse effects | continuously
Laboratory based toxicity | continuously
Adherence | continuously

CONTACTS AND LOCATIONS:
Overall Officials: Morris Schambelan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Walker UA, Venhoff N. Uridine in the prevention and treatment of NRTI-related mitochondrial toxicity. Antivir Ther. 2005;10 Suppl 2:M117-23. PMID 16152713
- [Background] Walker UA, Venhoff N, Koch EC, Olschewski M, Schneider J, Setzer B. Uridine abrogates mitochondrial toxicity related to nucleoside analogue reverse transcriptase inhibitors in HepG2 cells. Antivir Ther. 2003 Oct;8(5):463-70. PMID 14640394
- [Background] Sommadossi JP, Carlisle R, Schinazi RF, Zhou Z. Uridine reverses the toxicity of 3'-azido-3'-deoxythymidine in normal human granulocyte-macrophage progenitor cells in vitro without impairment of antiretroviral activity. Antimicrob Agents Chemother. 1988 Jul;32(7):997-1001. doi: 10.1128/AAC.32.7.997. PMID 3190201
- [Background] Keilbaugh SA, Hobbs GA, Simpson MV. Anti-human immunodeficiency virus type 1 therapy and peripheral neuropathy: prevention of 2',3'-dideoxycytidine toxicity in PC12 cells, a neuronal model, by uridine and pyruvate. Mol Pharmacol. 1993 Oct;44(4):702-6. PMID 8232219
- [Background] Banasch M, Goetze O, Knyhala K, Potthoff A, Schlottmann R, Kwiatek MA, Bulut K, Schmitz F, Schmidt WE, Brockmeyer NH. Uridine supplementation enhances hepatic mitochondrial function in thymidine-analogue treated HIV-infected patients. AIDS. 2006 Jul 13;20(11):1554-6. doi: 10.1097/01.aids.0000237373.38939.14. PMID 16847412
- [Background] Walker UA, Langmann P, Miehle N, Zilly M, Klinker H, Petschner F. Beneficial effects of oral uridine in mitochondrial toxicity. AIDS. 2004 Apr 30;18(7):1085-6. doi: 10.1097/00002030-200404300-00025. No abstract available. PMID 15096820